CLINICAL TRIAL: NCT06678100
Title: Prevalence and Care Partner Burden of Individuals With Alzheimer's Disease
Brief Title: Swallowing Impairments in Adults With and Without Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cara Donohue, Ph.D. CCC-SLP, Assistant Professor, Director of Medical Speech-Language Pathology, Vanderbilt University Medical Center
Other Study IDs: 241954; 25AARG-NTF-1369514 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Caregiver Burden; Healthy Aging; Dysphagia
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy community dwelling adults: Healthy adults ≥ 60 years old with no prior history of neurological or respiratory diseases, swallowing impairments, or history of head and neck surgery, cancer, or radiation to the head or neck will be enrolled in this study.
- Adults with Alzheimer's Disease and their caregivers: Adults with a diagnosis of Alzheimer's disease and their caregivers will be enrolled in this study.

SUMMARY:
This research study is investigating whether people with Alzheimer's disease (AD) experience more changes to swallowing than their healthy age-matched peers. The prevalence of swallowing impairments in moderate-severe AD is high (85-93%), yet little is known about how swallow function evolves throughout the disease course in people with AD. The overall objective of this study is to evaluate swallowing function in adults with and without Alzheimer's disease. The investigator will also be involving the primary caregivers of individuals with Alzheimer's that are enrolled in the study to better understand the impact of swallowing impairments on the primary caregivers of those with Alzheimer's Disease.

Healthy adults and individuals with Alzheimer's disease will:

* undergo tests of cough and swallow function
* undergo tests of grip and tongue strength
* complete questionnaires

Caregivers of individuals with Alzheimer's disease will also complete questionnaires.

DETAILED DESCRIPTION:
This study will involve one in-person research visit that will last approximately 1-1.5 hours and will consist of a screening, cough testing, swallow function testing, assessments of hand grip and tongue strength, and completion of questionnaires. Caregivers of those with Alzheimer's disease will also complete questionnaires.

ELIGIBILITY:
Inclusion criteria for AD cohort:

1. adult ≥60 years old
2. diagnosis of AD by a neurologist (confirmed with imaging, spinal tap, behavioral testing)
3. no prior history of other neurological diseases (aside from stroke which has resolved with no current symptoms)
4. no prior history of respiratory diseases
5. no prior history of head and neck surgery/head and neck cancer/radiation to head and neck region
6. consuming some form of oral intake
7. able to follow basic directions
8. able/willing to provide consent/assent.

Exclusion Criteria for AD Cohort:

1. individual <60 years old
2. Diagnosis of another type of dementia
3. History of neurological/respiratory diseases
4. History of head and neck surgery/head and neck cancer/radiation to head and neck region
5. not consuming any oral intake
6. Unable to follow basic directions
7. Unable to provide consent based on the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC), score <15 OR provide assent and a legal guardian provides consent.

Inclusion criteria for care partners of individuals with AD will be:

1. care partner of an individual with AD
2. willing to complete questionnaires/participate in an interview.

Exclusion Criteria for Caregivers of Individuals with AD:

1. not the primary caregiver of an individual with AD
2. unwilling to complete questionnaires/semi-structured interview

Inclusion criteria for community-dwelling adults will be:

1. adult ≥60 years old
2. no prior history of neurological diseases (aside from stroke which has resolved with no current symptoms)
3. no prior history of respiratory diseases

3) no prior history of head and neck surgery/head and neck cancer/radiation to head and neck region 4) no prior history of swallowing difficulties based on participant report. 5) Score ≥25th percentile based on sex/age/education/race on the Montreal Cognitive Assessment (MOCA)

Exclusion Criteria for Healthy Cohort:

1. individual <60 years old
2. history of neurological disease
3. history of respiratory disease
4. history of head and neck surgery/head and neck cancer/radiation to head and neck region
5. history of swallowing difficulties
6. Score <25th percentile based on sex/age/education/race on the Montreal Cognitive Assessment (MOCA)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The overall objective of this proposal is to evaluate swallow function in 80 healthy adults and 80 individuals with AD and to evaluate caregiver perceptions of swallow function and burden in 80 caregivers of individuals with AD. Thus, this study will enroll healthy adults, individuals with AD, and caregivers of individuals with AD.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Swallowing safety | During baseline visit at time of enrollment.
  The penetration aspiration scale is a validated 8-point ordinal rating scale that measures the depth of airway invasion and the patient's response during swallowing. Scores range from 1 to 8 with a score of 1 indicating a safe swallow (best score) and 8 indicating silent aspiration (worst score).

SECONDARY OUTCOMES:
Voluntary cough peak expiratory flow | During baseline visit at time of enrollment
  A measure of cough strength
Grip strength | During baseline visit at time of enrollment.
  Grip strength be used to quantify clinical frailty using a digital hand dynamometer.
Tongue strength | During baseline visit at time of enrollment.
  Tongue strength will be assessed using the Iowa Oral Pressure Instrument (IOPI).
Swallowing and Eating Related Fatigue Questionnaire (SERF) | During baseline visit at time of enrollment.
  Scores on the SERF range 0-48 with higher scores indicating greater impairment.
Swallowing Related Quality of Life Questionnaire (SWAL-QOL) | During baseline visit at time of enrollment.
  Scores on the SWAL-QOL range from 0-100 with lower scores indicating greater impairment.
Eating Assessment Tool 10 (EAT-10) | During baseline visit at time of enrollment.
  The EAT-10 contains 10 questions (score range: 0-40), higher scores indicate greater impairment.
Caregiver Analysis of Reported Experiences with Swallowing Disorders (CARES) Questionnaire | During baseline visit at time of enrollment.
  Scores on the CARES range from 0-26 with higher scores indicating greater caregiver burden.
Caregiver Self-Assessment Questionnaire | During baseline visit at time of enrollment.
  Scores range from 0-16 with higher scores indicating greater caregiver burden
3 oz water swallow test | During baseline visit at time of enrollment.
  Participants will be given a cup of three ounces of water and instructed to drink the water continuously. Fail criteria includes interrupted drinking and/or coughing/throat clearing during or immediately following the drinking task.
Reflex cough | During baseline visit at time of enrollment.
  Participants will undergo reflex cough testing.
Screening for Oral Frailty Tool (SOFT) | During baseline visit at time of enrollment.
  Oral frailty will be assessed as present/absent using the Screening for Oral Frailty Tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No